CLINICAL TRIAL: NCT03509922
Title: A Randomized, Dose-controlled, Open-label, Parallel, 2-treatment Group, Single Center, Pilot Study to Evaluate the Effectiveness of Sarpogrelate on Blood Hyperviscosity in the Patients With Peripheral Arterial Disease
Brief Title: A Study to Evaluate the Effect of Sarpogrelate on Blood Hyperviscosity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC036
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Peripheral Artery Disease, PAD
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — BID protein, human; sarpogrelate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anplag Tab. 100mg bid (Experimental): sarpogrelate hydrochloride 100mg bid for 24 weeks
  Interventions: Drug: Anplag Tab. 100mg bid
- Anplag Tab. 100mg tid (Experimental): sarpogrelate hydrochloride 100mg tid for 24 weeks
  Interventions: Drug: Anplag Tab. 100mg tid

INTERVENTIONS:
Drug: Anplag Tab. 100mg bid — sarpogrelate hydrochloride 100mg bid for 24 weeks
  Other Names: Sarpogrelate 200mg
  Arms: Anplag Tab. 100mg bid
Drug: Anplag Tab. 100mg tid — sarpogrelate hydrochloride 100mg tid for 24 weeks
  Other Names: Sarpogrelate 300mg
  Arms: Anplag Tab. 100mg tid

SUMMARY:
This study is to evaluate the effect of sarpogrelate on blood viscosity after 24 weeks in patients with high blood viscosity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with PAD* (*Criteria for diagnosis of PAD: diagnosed with Burger's disease, obstructive arteriosclerosis, diabetic peripheral vascular disease, or with ischemic symptoms such as ulcers, pain, cold sensation, etc.)
2. tODI < 3 at randomization
3. Aged ≥ 19 years
4. Written informed consent

Exclusion Criteria:

1. Patients requiring acute or two or more antiplatelet agents
2. Patients requiring anticoagulant therapy
3. Patients requiring surgical procedure due to vascular occlusion
4. Patients whose results are confirmed at the screening as follows:

   * hemoglobin (Hb) test value: male < 13 g/dL, female < 12 g/dL
   * platelet count < 60,000/µL
   * severe renal disease (eGFR < 30 mL/min/1.73 m2)
5. Patients with a history of cerebrovascular and cardiovascular complications (cerebral infarction, transient ischemic attack, myocardial infarction, unstable angina, coronary artery bypass, percutaneous coronary intervention) within the last 6 months
6. Contraindications stated in the SPC of sarpogrelate
7. Patients who are pregnant or planning to become pregnant
8. Those participating in other clinical trials with administration of investigational products at the screening
9. Those who are deemed to be ineligible to participate in the trial by investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 24 in tissue oxygen delivery index (tODI) | baseline, week 24

SECONDARY OUTCOMES:
Change from baseline to week 12 in tODI | baseline, week 12
Proportion of subjects with tODI elevated by 20% or more | baseline, week 12, week 24
Change from baseline to week 24 in 36-Item Short Form Health Survey (SF-36) | baseline, week 24

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Uijeongbu ST. Mary's Hospital, Uijeongbu-si, Gyeonggido, South Korea